CLINICAL TRIAL: NCT01707901
Title: A Randomised, Double-blind, Placebo-controlled, Two-period Crossover Study to Investigate the Effect of ONO-8539 on Oesophageal Pain Hypersensitivity in Patients With Non-erosive Reflux Disease
Brief Title: A Study of the Effect of ONO-8539 on Oesophageal Pain Hypersensitivity in Patients With Non-erosive Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-8539POE011
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: GERD
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ONO-8539

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONO-8539 (Experimental): ONO-8539
  Interventions: Drug: ONO-8539
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ONO-8539 — Treatment
  Other Names: Experimental
  Arms: ONO-8539
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A random controlled study to investigate the effect of a new drug, ONO-8539, on oesophageal pain hypersensitivity in patients with gastric reflux disease

DETAILED DESCRIPTION:
This is a Randomised, Double-blind, Placebo-controlled, Two-period Crossover Study to Investigate the Effect of ONO-8539 on Oesophageal Pain Hypersensitivity in Patients With Non-erosive Reflux Disease

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18-70 years inclusive with confirmed GERD and normal oesophageal mucosa will be enrolled in this study. Subjects demonstrate moderate intensity heartburn while being on a stable dose of proton pump inhibitor and demonstrate oesophageal hypersensitivity following distal oesophageal acid perfusion.

Exclusion Criteria:

* Subjects will be excluded if they have a motility disorder, are not able to tolerate study procedures or have had GI surgery or have a condition that would affect the study results. Subjects with functional heartburn, acute GI symptoms, endoscopic or manometric abnormality or a protocol-specified cardiovascular condition will not be enrolled.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of ONO-8539 on oesophageal pain hypersensitivity to acid perfusion | 28 Days
  Daily, through a pain assessment score chart

SECONDARY OUTCOMES:
To evaluate the effect of ONO-8539 on subject-reported symptoms of GERD | 28 Days
  Daily, by observation
To assess the tolerability of ONO-8539 | 28 Days
  Daily, through observation
To investigate the effect of ONO-8539 on oesophageal pain hypersensitivity to electrical stimulation | 28 Days
  Daily, through observation and a pain score chart
To evaluate the effect of ONO-8539 on quality of life | 28 Days
  Daily, through Quality of life assessment questionnaires
To investigate the pharmacokinetics of ONO-8539 | 28 Days
  AUC, Cmax, Tmax
  Concentrations of ONO-8539
To investigate the association among the changes in pharmacodynamics of ONO-8539 | 28 Days
  Daily observation and through Quality of life assessment questionnaires
To investigate the association between the changes in pharmacodynamic parameters of ONO-8539 and the plasma concentrations of ONO-8539 | 28 Days
  Correlation between pharmacokinetic results and study specific procedure results
To evaluate the use of antacid in each treatment group | 28 Days
  Daily record of frequency of use
To assess the safety of ONO-8539 | 28 days
To investigate the association among the changes in psychological parameters of ONO-8539 | 28 days
  Psychological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Clinical Department, Ono Pharmaceutical Co. Ltd
Locations (2):
- Leuven Clinical site, Leuven, Leuven, Belgium
- London Clinical site, London, London, United Kingdom